CLINICAL TRIAL: NCT06231771
Title: A Randomized, Double Blind, Placebo Controlled, Phase I/II Study Assessing the Efficacy and Safety of Peri-Ulcer Administration of Wharton-Jelly Mesenchymal Stem Cells in Patients With Non-Healing Diabetic Foot Ulcer
Brief Title: Safety and Efficacy of Stem Cells for Diabetic Foot Ulcer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Supergenics Life Science Sdn. Bhd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGT-DFU-23-001
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Diabetic Foot Ulcer
Keywords: DFU; Stem cells; Per-ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Equipment and Supplies; Excipients; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Dosage · Dosing of IMP is based on ulcer size. The recommended dose is 1 million cells/cm2 of ulcer. Administration · Injections will be done through peri-ulcer route. · Injection will be done 0.75 cm from the edge of the ulcer. · Injection will be done using 24G. The volume of injection will 4.0 - 6.0 ml per patient (maximum 0.1 to 0.2 ml per injection; 30 injections maximum per patients) Dosage · Dosing of placebo is based on ulcer size. the volume will be same as the experimental groups which is 2 ml per 1cm2 Administration · Injections will be done through peri-ulcer route. · Injection will be done 0.75 cm from the edge of the ulcer. · Injection will be done using 24G. The volume of injection will 4.0 - 6.0 ml per patient (maximum 0.1 to 0.2 ml per injection; 30 injections maximum per patients)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allogeneic mesenchymal stem cells (MSCs) (Experimental): Peri-ulcer injection of Umbilical cord MSC (1.0 million cells/cm2 of the ulcer) will be administered at multiple sites (maximum of 30 sites) with intervals of 3 cm x 3 cm around the ulcer with total volume of 0.1 to 0.2 ml per injection. Whatever IMP is drawn into the syringe for administration to the wound must be completely dispensed and nothing should be left in the syringe. Number of injections and volume of each injection can be as per Investigator's discretion. The same to be recorded in the source notes and CRF.The injection will be done approximately using a 24G needle and 1 ml/3ml syringe approximately within 0.75 cm from the edge of the ulcer. The needle should enter the base of the ulcer from the edge. After injection, patients must be in a lying down position for at least one hour in daycare center at the site and monitoring of oxygen saturation will be done up to 2 hours ± 10 minutes after the administration of the product.
  Interventions: Drug: Allogeneic mesenchymal stem cells (MSCs)
- Normal Saline (Placebo Comparator): The blinded placebo group will be injected with normal saline (NSand the volume to be injected is similar to the area of ulcer (2 mL of normal saline per 1 cm2 of ulcer). each injection will be o.1 to 0.2 ml normal saline (maximum injection will be 30 injection peri ulcer)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Allogeneic mesenchymal stem cells (MSCs) — Dosage · Dosing of IMP is based on ulcer size. The recommended dose is 1 million cells/cm2 of ulcer. Administration · Injections will be done through peri-ulcer route. · Injection will be done 0.75 cm from the edge of the ulcer. · Injection will be done using 24G. The volume of injection will 4.0 - 6.0 ml per patient (maximum 0.1 to 0.2 ml per injection; 30 injections maximum per patients)
  Other Names: Ex-vivo cultured allogeneic mesenchymal stem cells (MSCs) supplied in vials consisting of 3 million cells, suspended in 1.5 ml saline.
  Arms: Allogeneic mesenchymal stem cells (MSCs)
Drug: Normal Saline — Dosage · Dosing of placebo is based on ulcer size. the volume will be samed as the experimental groups which is 2 ml per 1cm2 Administration · Injections will be done through peri-ulcer route. · Injection will be done 0.75 cm from the edge of the ulcer. · Injection will be done using 24G. The volume of injection will 4.0 - 6.0 ml per patient (maximum 0.1 to 0.2 ml per injection; 30 injections maximum per patients)
  Other Names: Placebo (Normal Saline)
  Arms: Normal Saline

SUMMARY:
The objective of this clinical trial is to evaluate the effectiveness and safety of Wharton-Jelly mesenchymal stem cells administered around the ulcer site in patients with nonhealing diabetic foot ulcers. The key inquiries it seeks to address include the percentage of patients achieving complete healing/closure of the specified ulcer at any point during the 6-week period, the duration required for the complete closure of the target ulcer, and the nature and occurrence of adverse events (AEs), along with the total number of AEs and the proportion of patients experiencing AEs.

Patients meeting the eligibility criteria will receive either allogeneic mesenchymal stromal cells (MSC) or a placebo. The peri-ulcer injection of umbilical cord MSC or placebo will be administered at multiple locations, around the ulcer. Subsequent follow-up after the administration of umbilical cord MSC or placebo will be conducted to monitor and observe the progress of ulcer healing.

DETAILED DESCRIPTION:
Research involving MSCs promises new treatments and possible cures for many chronic and debilitating diseases. It has been shown that MSCs could be an effective therapy for many diseases, including CLI, AMI, OA of the knee, LC and DFU. No significant side effects have been reported with allogeneic MSC therapy in preclinical and clinical studies. Also, the potential benefits of MSC technology are compelling and worthy of pursuit in accordance with the appropriate ethical standards and regulatory guidelines. Both basic and clinical research suggest that allogeneic MSCs are likely to solve many unmet clinical needs, and this can be made available as an off-the-shelf product. the injective if this study was to evaluate the efficacy of peri-ulcer administration of Umbilical cord MSC in the healing of DFU and assess the safety of peri-ulcer administration of Umbilical cord MSC in DFU by assess the • Proportion of patients with complete healing/closure of the target ulcer at any time during the 6-weeks period and proportion of patients with sustained complete closure for additional 6-weeks of follow-up. besides that, this study also will assess the time to complete closure of target ulcer and rate of reduction in the size of the target ulcer during the 6 weeks of follow-up and proportion of patients with at least 50% closure of target ulcer during the 6-weeks period. this study is Double-blind, placebo-controlled, randomized trial. Estimated duration for the main protocol (e.g., from starts of screening to last subject processed and end of the study) is approximately 9 months at Hospital Canselor Tunku Muhriz (HCTM), Jalan Yaacob Latif, Bandar Tun Razak, 56000 Kuala Lumpur, Wilayah Persekutuan, Malaysia using Ex-vivo cultured allogeneic mesenchymal stem cells (MSCs) supplied in vials consisting of 3 million cells, suspended in 1.5 ml saline (3 million cells/1.5 mL) with dosage of 1 million cells/cm2 of ulcer. The administration of the product will be through the peri-ulcer route. The injection will be done using a 24G needle and 1 ml/3 ml syringe approximately within 0.75 cm from the edge of the ulcer. The needle should enter the base of the ulcer from the edge.

Injection of Umbilical cord MSC (1 million cells/cm2 of the ulcer) will be administered at multiple sites (maximum of 30 sites) with intervals of 3 cm x 3 cm around the ulcer in a total volume of 0.1 to 0.2 ml per injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-70 years old.
* Patients have type 2 diabetes mellitus
* Patients with HbA1c, less than or equal to 10%.
* Patients who were presented with an ulcer size between 8 to 12 cm2, have been diagnosed as full-thickness DFU.
* Adequate vascular perfusion (ABI ≥ 0.7 and < 1.3)
* Patients who are able and willing to provide consent and agree to comply with study procedures and follow-up evaluations.

Exclusion Criteria:

* Patients who are not diabetic.
* Patients with 2 or more ulcers.
* Patients with a history of participating in another stem cells trial or therapy within 3 months.
* Patients who are unsuitable to participate the clinical trial as determined by Investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with complete healing/closure of the target ulcer at any time during the 6-weeks period. | The monitoring of ulcer healing progress will continue until week 6 after the administration of the investigational medicinal product (IMP). The primary measure of effectiveness will be evaluated during the 8th visit which will take place at week 6.
  ulcer assessment (area and photograph)

SECONDARY OUTCOMES:
The proportion of patients with sustained complete closure for additional 6-weeks of follow-up. | weekly follow up 4 times, followed by biweekly followed up two times and one monthly follow up (weeks 12)
  ulcer assessment (area and photograph)
Time to complete closure of target ulcer. | weekly follow up 4 times, followed by biweekly followed up two times and one monthly follow up (weeks 12)
  ulcer assessment (area and photograph)
Rate of reduction in the size of the target ulcer during the 6 weeks of follow-up. | weekly follow up 4 times, followed by biweekly followed up two times and one monthly follow up (weeks 12)
  ulcer assessment (area and photograph)
The proportion of patients with at least 50% closure of target ulcer during the 6-weeks period | weekly follow up 4 times, followed by biweekly followed up two times and one monthly follow up (weeks 12)
  ulcer assessment (area and photograph)

CONTACTS AND LOCATIONS:
Overall Officials: Mohd Yazid Bajuri, Principal Investigator — Hospital Canselor Tunku Muhriz (HCTM)